CLINICAL TRIAL: NCT06709599
Title: Temporal Dynamics of Biochemical and Psychological Markers of Fatigue and Recovery in Mixed Martial Arts Athletes Undergoing Strength and Conditioning Training
Brief Title: Dynamics of Fatigue and Recovery in MMA Training
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Joanna Ostapiuk-Karolczuk, Principal Investigator, Poznan University of Physical Education
Other Study IDs: MMA546/11
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Athletes; Training; Fatigue; Recovery
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MMA athletes: Healthy, trained athletes
  Interventions: Other: Three-Week Strength and Conditioning Program

INTERVENTIONS:
Other: Three-Week Strength and Conditioning Program — Athletes train six days a week for three weeks, totaling approximately 15 hours of training per week. Training includes circuit training, weightlifting, technique drills, and sparring, designed to mimic typical MMA preparation.

SUMMARY:
This observational study aims to understand how strength and conditioning training impacts biochemical and psychological markers of fatigue and recovery in mixed martial arts (MMA) athletes. The main questions it aims to answer are:

How does a high-intensity training program affect key biochemical markers, such as cortisol, inflammation, and muscle damage indicators? How does this training influence psychological factors, such as stress, mood, and recovery states? Researchers will compare measurements taken at four time points during the study to see if the training program leads to changes in these markers and whether it effectively balances stress and recovery.

Participants will:

Undergo a structured strength and conditioning program for three weeks. Provide blood samples for biochemical analysis at four different times. Complete psychological questionnaires assessing mood, stress, and recovery states.

The findings aim to help optimize training programs and improve athlete well-being while minimizing the risk of overtraining.

DETAILED DESCRIPTION:
This study investigates the physiological and psychological responses of mixed martial arts (MMA) athletes to a structured high-intensity strength and conditioning training program. The primary focus is on monitoring temporal changes in key biochemical markers (e.g., cortisol, catecholamines, inflammatory cytokines) and psychological factors (e.g., mood profiles, stress, recovery states) to understand the balance between training-induced fatigue and recovery.

The study is conducted over three weeks, during which athletes follow a standardized training regimen comprising strength, endurance, and technical drills. Training intensity and volume are carefully managed, with no changes introduced during the observation period to ensure consistent data collection. Baseline measurements are taken 48 hours after a rest period to eliminate the effects of prior workouts.

Key Features:

Biochemical Analysis:

Blood samples are collected at four time points (pre-study, and after each training week) under standardized conditions, including morning fasting to minimize variability due to circadian rhythms.

Markers such as cortisol, catecholamines, hs-CRP, myoglobin, and urea are analyzed using validated ELISA protocols and biochemical kits.

Psychological Assessment:

The RESTQ-76 SPORT (Recovery-Stress Questionnaire for Athletes) and POMS (Profile of Mood States) questionnaires are administered before each blood sample collection to evaluate athletes' stress-recovery balance and mood states.

Training Protocol:

Athletes train six days a week for approximately 15 hours total per week. Training includes a mix of circuit training, weightlifting, technique drills, and sparring, designed to mimic typical MMA preparation.

Study Goals:

This study aims to determine the effects of a high-intensity training regimen on the interaction between physiological stress markers and psychological states. It seeks to provide insights into early indicators of overtraining and inform personalized approaches to athlete training that optimize performance while reducing injury risk.

By integrating biochemical and psychological data, this research highlights the need for a holistic approach to training management in MMA athletes, with implications for broader sports science and athletic performance enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 5 years of training experience in mixed martial arts (MMA).
* Training at least three times per week.
* At least two years of competitive fighting experience.
* Not using anabolic steroids, nutritional supplements, or medications that could influence study results.
* Maintaining a balanced diet throughout the study.
* Non-smoker.

Exclusion Criteria:

* Presence of any injury or clinical condition preventing participation in the study.
* Use of anti-inflammatory drugs.
* Undergoing a weight-cutting period during the study.

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility to participate in the study was restricted to male participants only.
Study Population: The study population consisted of male mixed martial arts (MMA) athletes affiliated with a sports club, actively engaged in regular training. All participants had a minimum of five years of training experience and at least two years of competitive fighting experience. They trained at least three times per week, maintained a balanced diet throughout the study, and did not use anabolic steroids, nutritional supplements, or medications that could influence the study results. The study was conducted during a training program that was an integral part of their preparation for competition. Athletes with injuries, clinical conditions, or those undergoing weight-cutting periods were excluded to ensure homogeneity and reliability of the results.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09-06 (Actual); Primary Completion 2014-09-20 (Actual); Study Completion 2015-05-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in cortisol level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of stress level.
Changes from baseline in epinephrine level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of sympathetic nervous system activity
Changes from baseline in norepinephrine level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of sympathetic nervous system activity, indicating stress response.
Changes from baseline in testosterone level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of the anabolic processes level.
Changes from baseline in hs CRP level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker inflammatory response.
Changes from baseline in creatine kinase level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker muscle damage.
Changes from baseline in total protein level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of protein catabolism, and recovery processes.
Changes from baseline in urea level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of balance between protein breakdown and recovery.
Changes from baseline in uric acid level. | At rest (before training), after the first week of training, and after the second and third weeks of training
  Marker of oxidative stress and, purine metabolism.
Mood Profile of Athletes Before Exercise Test Using POMS Questionnaire. | At rest (before training), after the first week of training, and after the second and third weeks of training
  The Profile of Mood States (POMS) questionnaire measures mood states and emotional well-being.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available because protecting participant confidentiality is a priority, especially given the sensitive nature of personal health and performance data collected in this study. Additionally, there may be limitations in data-sharing infrastructure and resources needed to anonymize and securely manage IPD for external access. Ensuring compliance with privacy regulations and ethical standards also restricts the feasibility of making IPD broadly available to other researchers.